CLINICAL TRIAL: NCT05393791
Title: ANZadapt: Phase II Randomised Controlled Trial of Patient-specific Adaptive Versus Continuous Abiraterone or eNZalutamide in Metastatic Castration-resistant Prostate Cancer
Brief Title: Phase II Randomised Controlled Trial of Patient-specific Adaptive vs. Continuous Abiraterone or eNZalutamide in mCRPC
Acronym: ANZadapt
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Anticancer Fund, Belgium (Other)
Responsible Party: Principal Investigator, dr. Tom van der Hulle, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79835; ANZUP 2101 (Other: ANZUP)
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Antineoplastic Agents, Hormonal; Evolution; Quality of Life; Prostatic Neoplasms, Castration-Resistant / drug therapy
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Intervention Model Description: Control group and experimental group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the experimental group, treatment will be paused if there is a >50% decline in baseline PSA. AA/ENZ will be restarted if the PSA rises to the same level or higher than the pre-treatment PSA. AA/ENZ treatment will be paused again after the PSA declines >50% from the baseline. This pause/restart cycle of adaptive therapy will be repeated presuming consent, tolerance and safety. Patients who do not have a >50% decline of their baseline PSA level after restarting AA/ENZ remain on treatment until the criteria for treatment failure are met.
  Interventions: Other: Patient-specific adaptive therapy; Drug: Abiraterone acetate; Drug: Enzalutamide
- Control group (Active Comparator): In the control group, patients will receive the standard continuous treatment with abiraterone or enzalutamide (AA/ENZ) until criteria for treatment failure are met.
  Interventions: Drug: Abiraterone acetate; Drug: Enzalutamide

INTERVENTIONS:
Other: Patient-specific adaptive therapy — Patients will start taking abiraterone or enzalutamide (AA/ENZ) daily. PSA will be measured every month as well as radiological evaluation by CT-scan and bone scan. Treatment will be continued until PSA has dropped >50%. The treatment will then be paused. Once the PSA has risen again above the pretreatment baseline, treatment will be re-initiated. AA/ENZ will be stopped again after the PSA declines >50% from the baseline. This will be continued until criteria for treatment failure are met (death by any cause or at least 2 out of 3 of the following events while on treatment: radiographic progression on CT-scan and/or bone scan, PSA progression or clinical progression).
  Arms: Experimental group
Drug: Abiraterone acetate — Use of abiraterone or enzalutamide
  Other Names: Zytiga
Drug: Enzalutamide — Use of abiraterone or enzalutamide
  Other Names: Xtandi

SUMMARY:
Hormone tablets, abiraterone (Zytiga®) and enzalutamide (Xtandi®) are approved to treat advanced prostate cancer. However, even if these drugs are helpful, their effectiveness usually diminishes over time. Small pilot studies have indicated that using hormone tablets sparingly, for just long enough to control the cancer, followed by a break in treatment and restarting them later, seems to improve how long hormone tablets can control the cancer. This study aims to find out if this pause/restart strategy is better than taking hormone tablets every day continuously. The study will include 168 people with metastatic castrate resistant prostate cancer in the Netherlands and Australia. Patients will be randomly 1:1 assigned between the control group and the experimental group. In the control group, patients will take the treatment with AA/ENZ every day until the prostate cancer doesn't respond anymore to the treatment. In the experimental group, patients will start with daily AA/ENZ until the PSA has declined for >50%. The treatment will then be paused and monthly PSA measurements will be performed. The treatment will be re-initiated when the PSA has increased to the level of before starting treatment. The treatment will be continued daily until the PSA has again dropped for >50%. This pause/restart cycle will be repeated until the prostate cancer doesn't respond anymore to the treatment.

DETAILED DESCRIPTION:
Abiraterone and enzalutamide (AA/ENZ) are drugs which are being used to treat metastatic prostate cancer. These drugs are a form of additional hormonal therapy and have been used for many years. For most patients, these drugs work well and the prostate cancer stays under control for several months to years. In all patients, there will be a moment when the prostate cancer doesn't respond anymore to the treatment. This is called resistance. This leads to increasement of PSA, tumor growth on the CT-scan and/or bone scan or decline of condition. The investigators want to establish if it is possible to delay the development of resistance by using the drugs differently. It is now recommended to use AA/ENZ daily until the prostate cancer doesn't respond anymore to the treatment. During treatment, all cancer cells sensitive to treatment will die and all cells resistant for treatment will survive. Based on evolutionary principles, this might not be a wise strategy. The groups of resistant cancer cells will prevail and will grow faster and faster. This will lead to increasement of PSA, tumor growth on the CT-scan and/or bone scan or decline of condition. The investigators want to establish if it is better to not take the treatment drugs daily, but to pause the treatment on regular basis. The theory of the investigators is that, due to just in time pausing the treatment, a part of the treatment sensitive cells will remain alive. These treatment sensitive cancer cells will compete with the treatment resistant cells for limited space and nutrients. In this way, the treatment sensitive cancer cells prevent the accelerating growth of the treatment resistant cancer cells. Due to this phenomenon, the investigator hypothesis is the prostate cancer will respond longer to treatment. It will take longer until a new treatment is necessary or until a patients develops complaints. When the treatment is paused, patients might experience less side effects. It is easy to establish whether the prostate cancer responds to treatment by measuring PSA.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent;
2. Aged 18 or older;
3. Histologically or cytologically confirmed adenocarcinoma of the prostate;
4. Ongoing androgen deprivation therapy with a GnRH analogue or bilateral orchiectomy (i.e. surgical or medical castration with testosterone at screening ≤1.7 nmol/L (<0.5 ng/mL)); patients who have not had a bilateral orchiectomy, must have a plan to maintain effective GnRH-analogue therapy for the duration of the trial;
5. Presence of metastatic disease on WBBS and/or CT-scan;
6. Progressive disease at study entry defined as per PCWG3 as one or more of the following criteria that occurred while the patient was on ADT:

   1. PSA progression defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each determination. Patients who received an anti-androgen must have progression after withdrawal (≥4 weeks since last flutamide or ≥6 weeks since last bicalutamide or nilutamide); OR
   2. Radiographic PD on bone scintigraphy and/or CT-scan;
7. A PSA concentration of ≥2 ng/mL.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
9. Controlled symptoms (opioids for cancer related pain stable for >4 weeks, no need for urgent radiotherapy for symptomatic lesions);
10. Estimated life expectancy of ≥12 months;
11. Patient has archival prostate cancer tissue available and which he consents to share or is willing to undergo a new tumour biopsy;
12. Adequate organ function: absolute neutrophil count > 1,500/μL (> 1.5*109/L); platelet count > 100,000/μL (> 100*109/L), haemoglobin > 90 g/L; total bilirubin < 1.5 times ULN, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 times ULN; creatinine < 175 μmol/L; albumin > 30 g/L;
13. Any other therapies for CRPC (excluding denosumab and bisphosphonates) have to be discontinued 3 weeks prior to study randomisation;
14. Able to swallow the study drug and comply with study requirements.

Exclusion Criteria:

1. Life-threatening or serious medical or psychiatric illness that could, in investigator's opinion, potentially interfere with participation in this study;
2. Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs. Potential participants with non-melanoma skin cancer, non-muscle invasive bladder cancer, or carcinoma in situ of any type are allowed if they have undergone complete resection;
3. Known or suspected brain metastasis or leptomeningeal disease;
4. Small-cell or neuroendocrine differentiation of prostate cancer;
5. Radiation therapy for treatment of the primary tumour within 3 weeks of screening visit;
6. Radiation or radionuclide therapy for treatment of metastasis within 3 weeks of screening visit, excluding radiation to reduce pain symptoms;
7. History of uncontrolled seizures (if patient and investigator wish to choose treatment with enzalutamide)
8. Unstable symptomatic ischemic heart disease, ongoing arrhythmias or New York Heart Association (NYHA) Class III or IV heart failure;
9. Known HIV infection, active chronic hepatitis B or C;
10. Known gastrointestinal (GI) disease that could interfere with GI absorption/tolerance of study drugs;
11. Prior treatments with CYP17 inhibitors (e.g. ketoconazole) or novel androgen receptor inhibitors (e.g. abiraterone, apalutamide, darolutamide or enzalutamide). Bicalutamide and nilutamide should be stopped >6 weeks before screening visit. Prior treatment with docetaxel in the mHSPC setting is allowed.
12. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As the investigated disease is prostate cancer, only males are eligible for inclusion.
Enrollment: 168 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | Time from randomization until death by any cause, or until criteria for treatment failure are met. PSA progression and clinical progression will be measured every 4 weeks, radiographic progression every 12 weeks, both up to 3 years after randomization.
  Defined as the time from randomization until death by any cause, or the occurrence of ≥2 of the following events:
  * Radiographic progression according to RECIST 1.1 and/or PWCG3 criteria on the CT-scan and/or WBBS while a subject received treatment with AA/ENZ during the whole period between the imaging tests. NB: Radiologic progression while a subject is off treatment in the experimental arm will trigger the endpoint, but may be an indication to restart treatment and continue with the adaptive dosing strategy
  * PSA progression, defined as an increase of PSA of >25% and >2 ng/mL occurring while a patient is on consecutive treatment with AA/ENZ for at least 8 weeks.
  * Clinical progression in the judgment of the treating clinician occurring while a patient is on consecutive treatment with AA/ENZ for at least 8 weeks.

SECONDARY OUTCOMES:
Time to PSA progression while on treatment | Time from randomization until an increase of PSA of >25% and >2 ng/mL persisting while a patient is on consecutive treatment for at least 8 weeks or death. PSA will be measured every 4 weeks until 3 years after randomization.
  defined as the time from randomization until an increase of PSA of >25% and >2 ng/mL persisting while a patient is on consecutive treatment for at least 8 weeks (according to PCWG3 criteria) or death. Patients without documented PSA progression or have not died will be censored at the last known time that the patient was progression-free. Patients who are lost to follow up will be censored at their last assessment time. Patients who begin a new anticancer treatment and have not had documented PSA progression will be censored at their last assessment point prior to beginning their new treatment.
Radiographic progression-free survival while on study treatment | Time from randomization to death or the first occurrence of radiographic progression while a subject received treatment between the imaging tests. Bone scan and CT-scan will be measured every 12 weeks until 3 years after randomization.
  Defined as the time from randomisation to first occurrence of radiographic progression by PCWG3 criteria and/or RECIST 1.1 on the CT-scan and/or WBBS while a subject received treatment with AA/ENZ during the whole period between the imaging tests or death. Patients without documented disease progression or have not died will be censored at the last known time that the patient was progression-free. Patients who are lost to follow up will be censored at their last assessment time. Patients who begin a new anticancer treatment and have not had a documented treatment failure event will be censored at their last assessment point prior to beginning their new treatment.
Overall survival | Time from randomization to the date of death due to any cause. Measured every 4 weeks up to 3 years after randomizaton and after end of treatment visit every 6 months until 2 years after end of treatment visit.
  defined as the time from randomization to the date of death due to any cause. For patients with no documented death by the end of the study, OS will be censored on the last date the patient was known to be alive. Patients who are lost to follow up will be censored at their last assessment time. Patients who begin a new anticancer treatment and have not had a documented treatment failure event will be censored at their last assessment point prior to beginning their new treatment.
Time to first skeletal-related event | Time from randomization to first skeletal-related event or death. Bone scan and CT-scan will be measured every 12 weeks up to 3 years after randomization.
  Time from randomization to first skeletal-related event or death will be assessed. A skeletal-related event is defined as radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression, or change of anti-neoplastic therapy to treat bone pain. Patients without documented skeletal-related event or have not died will be censored at the last known time that the patient was progression-free. Patients who are lost to follow up will be censored at their last assessment time. Patients who begin a new anticancer treatment and have not had a documented treatment failure event will be censored at their last assessment point prior to beginning their new treatment.
Health Related Quality of Life - FACT-P | FACT-P questionnaire will be obtained every 12 weeks up to 3 years after randomization
  FACT-P Quality of Life questionnaire
Health Related Quality of Life - EQ-5D-5L | EQ-5D-5L questionnaire will be obtained every 12 weeks up to 3 years after randomization
  EQ-5D-5L questionnaire.
Health Related Quality of Life - Pain | Brief Pain Inventory questionnaire will be obtained every 12 weeks up to 3 years after randomization
  Pain score per Brief Pain Inventory.
Adverse events | Adverse events will be measured every 12 weeks, up to 3 years after randomization.
  An adverse event is defined as any symptom, sign, illness, or untoward experience (including a clinically significant laboratory finding classified as Grade 3 or higher by the National Cancer Institute's Common Terminology Criteria for Adverse Events v5.0) that develops or worsens during the course of the study, whether or not the event is considered related to study drug. Such an event should be recorded as an adverse event only after the first dose of study drug is taken. Adverse events will be assessed every 12 weeks.

OTHER OUTCOMES:
Cost-effectiveness analysis | QoL and adverse events will be measured every 12 weeks up to 3 years after randomization. Treatment duration will be evaluated every 4 weeks up to 3 years after randomization.
  A cost-utility analysis will be performed from a healthcare perspective. Medication and other hospital costs will be assessed from hospital registrations. Quality-adjusted life years (QALYs) will be estimated using the Dutch tariff for the EQ-5D-5L (and the EQ-VAS as secondary analysis). Costs and QALYs will be extrapolated to a life-long horizon.
Cumulative duration on treatment | Every 4 weeks up to 3 years after randomization
  defined as the number of weeks on active treatment from randomization to the occurrence of treatment failure while on treatment.
Translational Biospecimens | Baseline and every 12 weeks
  Plasma samples suitable for circulating tumour DNA (ctDNA) analyses will be collected. The aim would be to perform explorative analyses on ctDNA to understand mechanisms of resistance, predictors of occurrence of progressive disease, and whether these results support the eco-evolutionary dynamics theory.

CONTACTS AND LOCATIONS:
Overall Officials: Tom van der Hulle, MD, Principal Investigator — Leiden University Medical Center; A/Prof. Craig Gedye, MBChB,FRACP, Study Chair — Australian and New Zealand Urogenital and Prostate Cancer Trials Group; Dr. Laurence Krieger, MBChB,FRACP, Principal Investigator — Australian and New Zealand Urogenital and Prostate Cancer Trials Group; Dr. Amy Rieborn, Principal Investigator — Leiden University Medical Center
Locations (19):
- Australia (12):
  - Border Medical Oncology Research Unit / The Border Cancer Hospital, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Genesis Care North Shore, St Leonards, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - ICON Cancer Centre, Adelaide, South Australia
  - Eastern Health Box Hill, Box Hill, Victoria
  - Fiona Stanly Hospital, Murdoch, Western Australia
- Netherlands (7):
  - Radboud Univeristy Medical Centre, Nijmegen, Gelderland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Isala Ziekenhuis, Zwolle, Overijssel
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Meander Medical Centre, Amersfoort, Utrecht
  - University Medical Center Groningen, Groningen